CLINICAL TRIAL: NCT04567589
Title: A Cross-sectional Study Among Healthcare Professionals in Canada to Assess Awareness and Knowledge of the Fibristal Additional Risk Minimization Measures
Brief Title: A Study to Evaluate Awareness and Knowledge of the Fibristal Additional Risk Minimization Measures Among Healthcare Professionals in Canada
Status: Withdrawn | Type: Observational
Why Stopped: This study was cancelled before any data collection due to business reasons.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-EPI-WH-0618
Record Dates: First submitted 2020-09-01; First posted 2020-09-28 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, cross-sectional survey study to evaluate the effectiveness of the Additional Risk Minimization Measures for Fibristal among Healthcare Professionals (HCPs).

DETAILED DESCRIPTION:
Data will be collected via web-based data capture by HCPs submitting surveys. The survey will be conducted in a single wave over 6 months. All data will be maintained in compliance with local regulations.

ELIGIBILITY:
Inclusion Criteria:

* HCPs have prescribed Fibristal for the indication of uterine fibroids within the past 6 months.
* HCPs have provided permission to share their responses in aggregate to Health Canada.

Exclusion Criteria:

* HCPs who participated in the cognitive pre-testing of the survey questionnaire to be used for the study.
* HCPs who have been direct employees of Allergan, ICON, Health Canada, or Professional Targeted Marketing (PTM) within the past 5 years.

Age Groups: Child, Adult, Older Adult
Study Population: The survey will endeavor to collect 150 completed HCP surveys.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of HCPs with correct responses to the knowledge level questions. | 18 - 24 months
  Correct responses to knowledge-related questions based on the contents of the Fibristal aRMMs.

SECONDARY OUTCOMES:
Percentage of HCPs that recall receiving and reading the HCP Letter and HCP Brochure . | 18 - 24 months
  HCP's recall of receiving and reading the HCP Letter and HCP Brochure .
Percenatage of HCPs that recall distributing the Fibristal Patient Alert Card | 18 - 24 months
  HCP's recall of distributing the Fibristal Patient Alert Card
Percentage of patients who recall counselling patients on information included in the Patient Alert Card | 18 - 24 months
  HCP's recall of counselling patients on information included in the Patient Alert Card
Overall score for each HCP will be calculated that totals the correct responses to all of the knowledge-related questions | 18 - 24 months
  Composite score on the level of HCPs knowledge across all knowledge-related questions.

CONTACTS AND LOCATIONS:
Overall Officials: Ahunna Ukah, Study Director — Allergan
Locations (1):
- Clinical Trials Registry Team, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/